CLINICAL TRIAL: NCT07135947
Title: To Evaluate the Clinical Impact of the Point Powered System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Point Designs (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Hanger Clinic: Prosthetics & Orthotics (Other); University of Colorado, Denver (Other); Infinite Biomedical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 348027; R44NS122687 (NIH)
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Amputation; Traumatic, Hand
Keywords: Prosthesis; Myoelectric; Digits; Fingers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Current/No Device (No Intervention): Baseline outcome measurements will be performed with subject's existing partial hand prosthetic treatment, as deemed standard-of-care by the patient's prosthetist. Device types include, but are not limited to, no prosthesis, passive prosthesis, passive positional prosthesis, body-powered prosthesis, myoelectric prosthesis, or other assistive device.
- Point Powered (Experimental): Outcome measurements will be performed after the subject has been fit with the Point Powered at 3 different points in time: immediately post-fitting, ~30 days post-fitting, and ~60 days post-fitting.
  Interventions: Device: Point Powered partial hand prosthetic system

INTERVENTIONS:
Device: Point Powered partial hand prosthetic system — The Point Powered system includes 1-4 3-joint mechatronic digits, low-profile EMG electrodes, a low-profile controller, and flexible batteries. These components will be integrated into a waterproof and dustproof packaging
  Arms: Point Powered

SUMMARY:
The objective of this study is to evaluate the efficacy of the Point Powered system as compared to the patient's standard-of-care treatment. This study will be a single subject crossover design where one group of 10 adult partial hand amputees will be evaluated on several metrics on their existing prosthetic treatment (Treatment 1) and the Point Powered system (Treatment 2) over a period of three months using standard two-site myoelectric control. Metrics include: in-clinic functional measures, subjective assessments, bilateral hand use, and prosthesis wear time.

ELIGIBILITY:
Inclusion Criteria:

* Partial unilateral hand loss with at least index and/or middle fingers amputated at the MCP level
* Intact thumb with full range of motion
* Fluent in English
* Age of 18 years or older

Exclusion Criteria:

* Patients with a residual limb that is unhealed from the amputation surgery
* Unhealed wounds
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Capacity for Myoelectric Control (ACMC) | Baseline (pre-fitting)
  The proctor for the measure chooses an everyday activity, such as setting up a table for snacks or replanting a flower, that is relevant to the study population. As the participants perform the chosen task, a trained rater will assess their capacity for control of their myoelectric prosthesis as represented by 30 items reflecting 6 aspects of quality of myoelectric control. These 6 aspects are "the need for external support," "grip force and opening width," "coordination of both hands, "in different positions and in motion (timing)," "repetitive grip and release," and "the need for visual feedback." Each item is scored on a 4-point scale and converted into linear measures of myoelectric control using Rasch analysis methods on the ACMC website. ACMC is the only measure that has been validated for individuals with upper limb (UL) loss who use myoelectric control and has been shown to demonstrate good test-retest reliability.
The Southampton Hand Assessment Procedure (SHAP) | Baseline (pre-fitting)
  The SHAP is a time based test of a standardized protocol of 26 timed activities of daily living (ADL) tasks. The SHAP has a set of "common objects" representative of everyday items for the user to pick up. The results of the SHAP is a score which directly compares the abilities of the subject with those of intact able-bodied individuals as well as more refined scores for six prehensile patterns. A SHAP score of 100 is what an intact person is expected to achieve. This test has been validated for normative data.
PROMIS Social Isolation | Baseline (pre-fitting)
  PROMIS Social Isolation is a self-reported person-centered measure that focuses on perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Ability to Participate | Baseline (pre-fitting)
  PROMIS Ability to Participate is a self-reported person-centered measure that focuses on perceived ability to perform one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Physical Function - Upper Extremity | Baseline (pre-fitting)
  PROMIS Physical Function - Upper Extremity is a self-reported person-centered measure that focuses on capability to perform activities that require use of the upper extremity including shoulder, arm, and hand. Examples include writing, using buttons, or opening containers. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Satisfaction with Social Roles and Activities | Baseline (pre-fitting)
  PROMIS Satisfaction with Social Roles and Activities is a self-reported person-centered measure that focuses on satisfaction with performing one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
Assessment of Capacity for Myoelectric Control (ACMC) | Immediately post-fitting
  The proctor for the measure chooses an everyday activity, such as setting up a table for snacks or replanting a flower, that is relevant to the study population. As the participants perform the chosen task, a trained rater will assess their capacity for control of their myoelectric prosthesis as represented by 30 items reflecting 6 aspects of quality of myoelectric control. These 6 aspects are "the need for external support," "grip force and opening width," "coordination of both hands, "in different positions and in motion (timing)," "repetitive grip and release," and "the need for visual feedback." Each item is scored on a 4-point scale and converted into linear measures of myoelectric control using Rasch analysis methods on the ACMC website. ACMC is the only measure that has been validated for individuals with upper limb (UL) loss who use myoelectric control and has been shown to demonstrate good test-retest reliability.
The Southampton Hand Assessment Procedure (SHAP) | Immediately post-fitting
  The SHAP is a time based test of a standardized protocol of 26 timed activities of daily living (ADL) tasks. The SHAP has a set of "common objects" representative of everyday items for the user to pick up. The results of the SHAP is a score which directly compares the abilities of the subject with those of intact able-bodied individuals as well as more refined scores for six prehensile patterns. A SHAP score of 100 is what an intact person is expected to achieve. This test has been validated for normative data.
PROMIS Social Isolation | Immediately post-fitting
  PROMIS Social Isolation is a self-reported person-centered measure that focuses on perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Ability to Participate | Immediately post-fitting
  PROMIS Ability to Participate is a self-reported person-centered measure that focuses on perceived ability to perform one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Physical Function - Upper Extremity | Immediately post-fitting
  PROMIS Physical Function - Upper Extremity is a self-reported person-centered measure that focuses on capability to perform activities that require use of the upper extremity including shoulder, arm, and hand. Examples include writing, using buttons, or opening containers. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Satisfaction with Social Roles and Activities | Immediately post-fitting
  PROMIS Satisfaction with Social Roles and Activities is a self-reported person-centered measure that focuses on satisfaction with performing one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
Assessment of Capacity for Myoelectric Control (ACMC) | 30 days post-fitting
  The proctor for the measure chooses an everyday activity, such as setting up a table for snacks or replanting a flower, that is relevant to the study population. As the participants perform the chosen task, a trained rater will assess their capacity for control of their myoelectric prosthesis as represented by 30 items reflecting 6 aspects of quality of myoelectric control. These 6 aspects are "the need for external support," "grip force and opening width," "coordination of both hands, "in different positions and in motion (timing)," "repetitive grip and release," and "the need for visual feedback." Each item is scored on a 4-point scale and converted into linear measures of myoelectric control using Rasch analysis methods on the ACMC website. ACMC is the only measure that has been validated for individuals with upper limb (UL) loss who use myoelectric control and has been shown to demonstrate good test-retest reliability.
The Southampton Hand Assessment Procedure (SHAP) | 30 days post-fitting
  The SHAP is a time based test of a standardized protocol of 26 timed activities of daily living (ADL) tasks. The SHAP has a set of "common objects" representative of everyday items for the user to pick up. The results of the SHAP is a score which directly compares the abilities of the subject with those of intact able-bodied individuals as well as more refined scores for six prehensile patterns. A SHAP score of 100 is what an intact person is expected to achieve. This test has been validated for normative data.
PROMIS Social Isolation | 30 days post-fitting
  PROMIS Social Isolation is a self-reported person-centered measure that focuses on perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Ability to Participate | 30 days post-fitting
  PROMIS Ability to Participate is a self-reported person-centered measure that focuses on perceived ability to perform one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Physical Function - Upper Extremity | 30 days post-fitting
  PROMIS Physical Function - Upper Extremity is a self-reported person-centered measure that focuses on capability to perform activities that require use of the upper extremity including shoulder, arm, and hand. Examples include writing, using buttons, or opening containers. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Satisfaction with Social Roles and Activities | 30 days post-fitting
  PROMIS Satisfaction with Social Roles and Activities is a self-reported person-centered measure that focuses on satisfaction with performing one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
Assessment of Capacity for Myoelectric Control (ACMC) | 60 days post-fitting
  The proctor for the measure chooses an everyday activity, such as setting up a table for snacks or replanting a flower, that is relevant to the study population. As the participants perform the chosen task, a trained rater will assess their capacity for control of their myoelectric prosthesis as represented by 30 items reflecting 6 aspects of quality of myoelectric control. These 6 aspects are "the need for external support," "grip force and opening width," "coordination of both hands, "in different positions and in motion (timing)," "repetitive grip and release," and "the need for visual feedback." Each item is scored on a 4-point scale and converted into linear measures of myoelectric control using Rasch analysis methods on the ACMC website. ACMC is the only measure that has been validated for individuals with upper limb (UL) loss who use myoelectric control and has been shown to demonstrate good test-retest reliability.
The Southampton Hand Assessment Procedure (SHAP) | 60 days post-fitting
  The SHAP is a time based test of a standardized protocol of 26 timed activities of daily living (ADL) tasks. The SHAP has a set of "common objects" representative of everyday items for the user to pick up. The results of the SHAP is a score which directly compares the abilities of the subject with those of intact able-bodied individuals as well as more refined scores for six prehensile patterns. A SHAP score of 100 is what an intact person is expected to achieve. This test has been validated for normative data.
PROMIS Social Isolation | 60 days post-fitting
  PROMIS Social Isolation is a self-reported person-centered measure that focuses on perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Ability to Participate | 60 days post-fitting
  PROMIS Ability to Participate is a self-reported person-centered measure that focuses on perceived ability to perform one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Physical Function - Upper Extremity | 60 days post-fitting
  PROMIS Physical Function - Upper Extremity is a self-reported person-centered measure that focuses on capability to perform activities that require use of the upper extremity including shoulder, arm, and hand. Examples include writing, using buttons, or opening containers. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.
PROMIS Satisfaction with Social Roles and Activities | 60 days post-fitting
  PROMIS Satisfaction with Social Roles and Activities is a self-reported person-centered measure that focuses on satisfaction with performing one's usual social roles and activities. Responses are scored on a scale of 1 to 5. Individual response scores are summed to get a raw score, which can be converted to a standardized T-score with a mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
Mean Prosthesis Wear Duration (MPWD) | Through study completion, an average of 3 months
  We will measure the mean duration of daily prosthesis wear as a proxy for improved prosthesis acceptance. Prosthesis wear time is defined as the time from when participants don their prostheses to the time they doff their prostheses. The time points are both recorded by participants and through analysis of the activity monitors. We believe the mean prosthesis wear duration is an important metric as it is possible that participants who have higher levels of satisfaction with their prosthesis will wear their prosthesis for long periods of time. It is also possible that wear time may not necessarily be correlated with corresponding usage of the prosthetic limb. Measuring this variable will be important in its assessment in comparison with other variables.
Bilateral magnitude (BM) | Through study completion, an average of 3 months
  Participants will be asked to wear accelerometers on each wrist throughout the study. From accelerometry data, we will calculate the bilateral magnitude (BM), which quantifies the intensity of activity across both arms for a given duration. A BM of 0 indicates that no activity occurs and increasing BMs indicate that more bilateral activity occurs.
Magnitude ratio (MR) | Through study completion, an average of 3 months
  Participants will be asked to wear accelerometers on each wrist throughout the study. From accelerometry data, we will calculate magnitude ratio (MR), which is the ratio of acceleration between the two arms for a given duration. A MR of 0 indicates equivalent contribution of activity from both arms; positive values of MR indicate that more prosthesis-side activity occurs and negative values of MR indicate that more sound-side activity occurs.
Secondary activity duration variables | Through study completion, an average of 3 months
  In addition to BM and MR, we will also calculate durations of non-injured UL activity, amputated UL activity, simultaneous UL activity, and total UL activity averaged across each day. Measurements of activity durations by UL side can provide additional insight into how much one side is used over another and with respect to bilateral use. This measure is complimentary to BM and MR measures and will help us determine if the Point Powered promotes more use of the prosthesis side relative to the standard-of-care.

CONTACTS AND LOCATIONS:
Overall Officials: Levin Sliker, PhD, Principal Investigator — Point Designs
Locations (3):
- United States (3):
  - University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado
  - Point Designs, Broomfield, Colorado
  - Hanger Clinic, Lafayette, Colorado

IPD SHARING:
Plan to Share IPD: No